CLINICAL TRIAL: NCT01602952
Title: A Phase I/II Multicenter Study of IY5511HCl in Philadelphia Chromosome Positive Chronic Myeloid Leukemia Patients Without Optimal Response or Tolerance to Bcr-Abl Tyrosine Kinase Inhibitors (Imatinib and/ or Dasatinib, Nilotinib)
Brief Title: Philadelphia Chromosome Positive CML Patients Without Optimal Response or Tolerance to Bcr-Abl TKI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IY5511A1201
Record Dates: First submitted 2012-04-20; First posted 2012-05-21 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Hematologic Diseases
Keywords: Radotinib; CML-CP, AP
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome; Hematologic Diseases | interventions — 4-methyl-N-(3-(4-methylimidazol-1-yl)-5-trifluoromethylphenyl)-3-(4-pyrazin-2-ylpyrimidin-2-ylamino)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radotinib (Experimental): Phase 1 : 200mg/kg or 1200mg/m^2
  Phase 2 : 400mg Bid
  Interventions: Drug: Radotinib

INTERVENTIONS:
Drug: Radotinib — 50mg, 100mg or 200mg Capsule BID
  Other Names: IY5511HCl

SUMMARY:
A Phase I/II multicenter study of IY5511HCl in Philadelphia chromosome positive chronic myeloid leukemia patients without optimal response or tolerance to Bcr-Abl tyrosine kinase inhibitors (Imatinib and/ or Dasatinib, Nilotinib) In this study, The efficacy and safety of CML patients who are resistant or intolerable to imatinib in the Chronic and Accelerated phases.

Phase 1

1. To investigate the Maximum Tolerated Dose (MTD) and the Dose Limiting Toxicity (DLT) of oral Radotinib HCl bid (twice daily) in the Philadelphia chromosome-positive CML subjects who are resistant, suboptimal responsive, or intolerant to imatinib OR resistant or intolerant to at least one second-generation targeted anticancer agent while being resistant, suboptimal responsive, or intolerant to imatinib simultaneously.

Phase 2

1. To investigate safety of oral Radotinib HCl in CML patients who are resistant or intolerable to imatinib in the chronic and accelerated phases.
2. To evaluate hematologic and cytogenetic efficacy of oral Radotinib HCl in CML patients who are resistant or intolerable to imatinib in the chronic and accelerated phases.

DETAILED DESCRIPTION:
This study is a multi-center, open-label, Phase 1/2 clinical trial of Radotinib HCl, a targeted anticancer agent that inhibits the Bcr-Abl oncoprotein. It is aimed at determining the optimal therapeutic dose and confirming safety and efficacy of Radotinib HCl. Phase 1 study began at St. Mary's hospital in Korea and Phase 2 study is ongoing at 9 Korean sites and about 7 sites in China, India and Thailand will take part in Phase 2. After determination of a safe and proper therapeutic dose in Phase 1, Phase 2 began continuously to evaluate efficacy in chronic and accelerated phases. Before the start of the Phase 2 trial, interim or final reports for the Phase 1 trial were reviewed by the Korean Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

Phase I

1. Age ≥ 18 years old
2. Ph+ CML patients who are resistant at chronic, accelerate, and acute phase, or suboptimal responsive, or intolerant to imatinib or resistant or intolerant to at least one second-generation targeted anticancer agent while being resistant, suboptimal responsive, or intolerant to imatinib simultaneously.
3. WHO Performance status of ≤2
4. Patients must have the following laboratory values With normal liver and renal function
5. Patients who have received interferon, other anti cancer drug or radiotherapy > 1 week prior to starting study drug.

Phase II

1. Age ≥ 18 years old
2. Ph+ CML patients in chronic or accelerated phase who are resistant or intolerant to Imatinib mesylate
3. WHO Performance status of ≤2
4. Patients must have the following laboratory values With normal liver and renal function
5. Patients who have received interferon, other anti cancer drug or radiotherapy > 1 week prior to starting study drug.

Exclusion Criteria:

Phase I

1. CNS infiltration
2. Impaired cardiac function, including any one of the followings.

   * LVEF <45% as determined by MUGA scan or echocardiogram
   * Clinically significant resting bradycardia
3. Severe GI disease that may cause drug absorption problem of study drug
4. Use of therapeutic Warfarin
5. Acute or chronic liver or renal disease
6. Other concurrent severe and/or uncontrolled medical conditions
7. Treatment with any hematopoietic colony-stimulating growth factors ≤1 week prior to starting study drug.
8. Patients who are currently receiving treatment with medications have the potential to prolong the QT interval
9. Patients who have received Imatinib, interferon, other anti cancer drug or chemotherapy ≤ 1 week
10. Patients who have received Nilotinib and Dasatinib ≤4 weeks prior to starting study drug.
11. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
12. Patients who are pregnant or breast-feeding or adults of reproductive potential not employing an effective method of birth control.
13. Patients not to agree using birth control during the study and for up 3 months following study completion.

15. HIV infection

Phase II

1. Blast phase CML
2. CNS infiltration
3. Impaired cardiac function, including any one of the following

   * LVEF< 45% as determined by MUGA scan or echocardiogram
   * Use of Cardiac pacemaker
   * ST depression > 1mm in 2 or more leads and/or T wave inversions in 2 or more contiguous leads
   * Congenital long QT syndrome
   * History of, or presence of significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia
   * QTcF> 480 msec on screening ECG
   * Right bundle branch block + left anterior hemiblock, Bifascicular block
   * Angina pectoris
4. Severe GI disease that may cause drug absorption problem of study
5. Use of therapeutic Warfarin
6. Acute or chronic liver or renal disease
7. Other concurrent severe and/or uncontrolled medical conditions
8. Treatment with any hematopoietic colony-stimulating growth factors ≤1 week prior to starting study drug.
9. Patients who are currently receiving treatment with medications have the potential to prolong the QT interval
10. Patients who have received Imatinib, interferon, other anti cancer drug or chemotherapy ≤ 1 week
11. Patients who have received wide field radiotherapy ≤4 weeks prior to starting study drug.
12. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
13. Patients who are pregnant or breast-feeding or adults of reproductive potential not employing an effective method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-07; Primary Completion 2012-10 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
To investigate the Maximum Tolerated Dose(Phase 1) | 12 month
  Radotinib will be given orally twice daily. Dose will be increased until it reaches MTD or the blood concentration of Radotinib stops rising
Rate of Complete hematologic response(CHR)(Phase 2) | 12 months
  Main parameters for response assessment in the chronic and accelerated phases include Major Hematologic Responses (MR; No Evidence of Leukemia or NEL + Complete Hematologic Response or CHR) lasting for 4 weeks and at least one major cytogenetic response (MCyR)

SECONDARY OUTCOMES:
To investigate the Dose Limiting Toxicity(Phase 1) | 12 months
  The initial cohort will include 3 subjects who will receive 100mg Radotinib daily. If DLT is observed in one of the 3 subjects, the same dose will be given to 3 more subjects to evaluate safety.
Rate of complete Cytogenetic Response(CCyR)(Phase 2) | 12 months
  Cytogenetic response rate will be calculated as the percentage of Ph+ bone marrow metaphases as follows at least 20 bone marrow metaphases should be analyzed.
Adverse events(Phase 1& Phase 2) | 12 months
  All adverse events recorded during the study will be itemized and summarized. Severity, relation to the study medication, and seriousness will be summarized for each adverse event.
Progression-free survival or PFS | 12 months
  It is defined as the duration from the first day of administration to the earliest day of disease progression or death for certain causes. In subjects who have shown response, disease progression is defined as loss of MCyR.

CONTACTS AND LOCATIONS:
Overall Officials: IL-yang Pharm, Study Director — IL-YANG Pharmaceutical.Co.,Ltd.
Locations (12):
- India (2):
  - Local institution, Mumbai, Maharashtra
  - Local institution, Mumbai, Mazagaon
- South Korea (9):
  - Local institution, Daegu, Buk-gu
  - Local institution, Jeonju, Deokjin-gu
  - Local institution, Ulsan, Dong-gu
  - Local institution, Anyang-si, Dongan-gu
  - Local institution, Hwasun, Hwasun-eup
  - Local institution, Seoul, Jongro-ku
  - Local institution, Busan, Seo-gu
  - Seoul St. Mary's hospital, Seoul, Seocho-gu
  - Local institution, Suwon, Yeongtong-gu
- Local institution, Bangkok, Phyathai, Thailand

REFERENCES:
- [Derived] Kim SH, Menon H, Jootar S, Saikia T, Kwak JY, Sohn SK, Park JS, Jeong SH, Kim HJ, Kim YK, Oh SJ, Kim H, Zang DY, Chung JS, Shin HJ, Do YR, Kim JA, Kim DY, Choi CW, Park S, Park HL, Lee GY, Cho DJ, Shin JS, Kim DW. Efficacy and safety of radotinib in chronic phase chronic myeloid leukemia patients with resistance or intolerance to BCR-ABL1 tyrosine kinase inhibitors. Haematologica. 2014 Jul;99(7):1191-6. doi: 10.3324/haematol.2013.096776. Epub 2014 Apr 4. PMID 24705186